CLINICAL TRIAL: NCT03943901
Title: A Phase II Study of Split-Dose R-CHOP in Older Adults With Diffuse Large B-cell Lymphoma
Brief Title: Split-Dose R-CHOP for Older Adults With DLBCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0138; 2019-0138 (Other: Institutional Review Board); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); A534260 (Other: UW Madison); Protocol Version 7/21/2023 (Other: UW Madison); NCI-2020-01530 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma; DLBCL; Cancer
Keywords: chemotherapy; cancer; elderly; lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Neoplasms; Lymphoma | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Split Dose R-CHOP (Experimental): Each cycle is 28 days and consists of one "A" treatment on Day 1 and one "B" treatment on Day 15 for 6 cycles
  Day 1 ("A" part of cycle)
  * Rituximab 375 mg/m2 IV (or biosimilars Ruxience or Truxima)
  * Cyclophosphamide 375 mg/m2 IV
  * Doxorubicin 25 mg/m2 IV
  * Vincristine 1 mg IV
  * Prednisone 50 mg (Days 1-5) PO
  * Pegfilgrastim (supportive care) 6 mg on Day 2 (24 hours after completion of chemotherapy) or filgrastim daily as institutionally indicated (starting 24 hours post completion of chemotherapy), or institutional standard granulocyte stimulating factor.
  Day 15 ("B" part of cycle)
  * Cyclophosphamide 375 mg/m2 IV
  * Doxorubicin 25 mg/m2 IV
  * Vincristine 1 mg IV
  * Prednisone 50 mg (Days 15-19) PO
  * Pegfilgrastim (supportive care) 6 mg on Day 16 (24 hours after completion of chemotherapy) or filgrastim daily as institutionally indicated (starting 24 hours post completion of chemotherapy), or institutional standard granulocyte stimulating factor.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Biological: Pegfilgrastim

INTERVENTIONS:
Drug: Rituximab — Rituximab is a monoclonal antibody
  Other Names: Rituxan
Drug: Cyclophosphamide — Chemotherapy drug, alkylating agent
  Other Names: Cytoxan
Drug: Doxorubicin — Chemotherapy drug, anthracycline antibiotic
  Other Names: Adriamycin
Drug: Vincristine — Chemotherapy drug, plant alkaloid
Drug: Prednisone — Steroid, anti-inflammatory
Biological: Pegfilgrastim — Granulocyte stimulating factor, biologic response modifier
  Other Names: filgrastim

SUMMARY:
This study is investigating a new administration schedule of Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (R-CHOP) chemotherapy for participants with Diffuse Large B-Cell Lymphoma (DLBCL), focusing on an underserved elderly population (aged 75 and up; certain participants 70-74 may be eligible) that is often excluded from clinical trials. Participants can expect to be on study for 2.5 years (treatment for 6 months and 2 years of post treatment follow-up).

DETAILED DESCRIPTION:
This study will test the efficacy of split-dose R-CHOP for the treatment of elderly patients with de novo diagnosis of DLBCL or transformed DLBCL. Split-dose R-CHOP involves giving Cyclophosphamide, Doxorubicin, Vincristine, Prednisone (CHOP) chemotherapy at 14 days' interval with Rituximab given once/month. The safety for every 14-day CHOP administration was studied in a large prospective randomized control trial of patients up to the age of 80 years. In this study, R-CHOP given every 14 days for up to 6 cycles was felt to be the best method of delivery of chemotherapy. Receiving greater than 6 cycles of R-CHOP chemotherapy was not found to be beneficial compared to participants receiving 6 cycles of R-CHOP. Additionally, an interim response adapted approach by combining imaging and MRD testing will be used to identify participants who will receive an abbreviated chemotherapy course if they are both Positron Emission Tomography/Computed Tomography (PET/CT) and Minimum Residual Dose (MRD) negative.

In the proposed study, participants will receive a 50% dose reduction of CHOP chemotherapy on Day 1 and Day 15 of each cycle with full dose Rituximab on Day 1 for up to a total of 6 months of chemotherapy. Participants who are MRD and PET/CT negative after 2 months will be placed on an abbreviated regimen with R-CHOP x 4 additional doses with full dose Rituximab and a 50% dose reduction in CHOP chemotherapy. The hypothesis is that this method of administration of R-CHOP will be a safe and effective form of chemotherapy for older patients with DLBCL and will allow older patients to receive curative intent treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent document indicating that the participant (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* All patients age ≥75 years and participants aged 70-74 years who are determined to be unfit or frail by Cumulative Illness Rating Score-Geriatrics (CIRS-G) scale

  * For participants aged 70-74 years: CIRS-G score with 5-8 comorbid conditions scored 2 or ≥1 comorbidity scored 3-4. CIRS-G score is to be reviewed by the study PI prior to enrollment.
* Newly diagnosed, untreated, biopsy proven CD20 positive DLBCL (including high grade B-cell lymphoma & T-cell/histiocytic rich large B-cell lymphoma). Participants with discordant bone marrow (i.e. involved by low-grade/indolent NHL) are eligible. Participants with transformed DLBCL from underlying low-grade disease are eligible. Participants with composite DLBCL and concurrent low-grade lymphoma are eligible.

  * Copy of pathology report must be sent to coordinating site to confirm diagnosis for eligibility
  * Participants with prior treatment for low grade NHL with non-anthracycline based regimens are eligible
* Measurable disease by PET/CT or Bone Marrow (BM) biopsy prior to enrollment
* Left ventricular ejection fraction ≥50% by resting echocardiography or resting Multi-gated acquisition (MUGA) scan
* Karnofsky Performance Score ≥50
* Ann Arbor Stage II bulky, III, or IV disease
* Minimum life expectancy greater than 3 months
* Negative HIV test
* For participants with hepatitis B virus antigen (HbsAg) or core antibody (HbcAb) seropositivity, participants must have a negative Hep B viral load and an appropriate prophylaxis plan must be in place during chemotherapy therapy treatment. For all participants that have Hep B core antibody positive, they should take entecavir prophylaxis (0.5 mg PO daily) until 1 year from completion of chemotherapy. Hep B viral load should be checked on these participants prior to starting chemotherapy and every 3 months thereafter if initial Hep B viral load is negative (+/- 1 week if chemotherapy cycle is delayed). If Hep B viral load is positive, Hepatology or Identification (ID) referral is recommended, and hepatitis B virus (HBV) viral load should be checked monthly
* For participants with hepatitis C Ab (HbcAb) positivity, a viral load must be checked and be negative for enrollment
* Intrathecal chemotherapy for central nervous system prophylaxis only can be given at the discretion of the primary oncologist

Exclusion Criteria:

* History of previous anthracycline exposure
* Central Nervous System (CNS) or meningeal involvement at diagnosis
* Creatinine Clearance <25 mL/min by body surface area (BSA)-adjusted Cockroft-Gault
* Poor hepatic function, defined as total bilirubin concentration greater than 3.0 mg/dL or transaminases over 4 times the maximum normal concentration, unless these abnormalities are felt to be related to the lymphoma.
* Pulmonary dysfunction defined as >2 L of oxygen required by nasal cannula to maintain peripheral capillary oxygen saturation (SpO2) ≥90% unless felt to be related to underlying lymphoma.
* Myocardial Infarction within 6 months of enrollment
* Active, uncontrolled infectious disease
* Known concurrent bone marrow malignancies (e.g. myelodysplastic syndrome) or poor bone-marrow reserve, defined as neutrophil count less than 1.5×10⁹/L or platelet count less than 100×10⁹/L, unless caused by bone-marrow infiltration with lymphoma
* History of a second concurrent active malignancy or prior malignancy which required chemotherapy treatment within the preceding 2 years
* Treatment with any investigational drug within 30 days before the planned first cycle of chemotherapy
* Unable or unwilling to sign consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2027-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Fletcher, MD, Principal Investigator — University of Wisconsin, Madison; Nirav Shah, MD, MS, Study Chair — Medical College of Wisconsin Clinical Cancer Center
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Split Dose R-CHOP
Started | 27
On Treatment | 26
Off Treatment | 26
Completed | 14
Not Completed | 13
Not completed — On Follow Up | 12
Not completed — deemed not eligible prior to starting treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Split Dose R-CHOP
Number analyzed (Participants) | 27
Age, Customized [Count of Participants; unit: Participants]
  70-79 years | 13
  80-89 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR)
Description: Simon 2-stage design with complete response (CR) rate at the end of treatment as our primary outcome. 40% is an unacceptable boundary for complete response rate and 60% as an acceptable complete response rate. CR at the end of treatment, will be estimated as the observed proportion and presented with a 95% Wilson confidence interval.
Time Frame: up to 6 months
Population: number of participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Split Dose R-CHOP
Number analyzed (Participants) | 26
Participants | 17

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS measures survival without relapse/progression or death starting from study enrollment. Relapse or progression of disease and death will be considered as events; subjects who survive without recurrence or progression will be censored at last contact. PFS will be estimated using the Kaplan Meier estimate and presented with graphically with pointwise 95% confidence intervals.
Time Frame: up to 2 years 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival (OS)
Description: OS measures time to death starting from study enrollment. Death from any cause will be considered an event; surviving subjects will be censored at time of last follow-up. OS will be estimated using the Kaplan-Meier estimate and presented with graphically with pointwise 95% confidence intervals. Exploratory Cox proportional hazards regression will be used to evaluate the effect of baseline covariates on PFS and OS.
Time Frame: up to 2 years 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Treatment Emergent Serious Adverse Events
Description: The incidence of serious adverse events will be reported for all subjects who received at least one dose of the study treatment. The proportion of subjects experiencing a Serious Adverse Event (SAE) will be reported with 95% confidence intervals overall. Toxicity will be monitored using the formal boundary described in the protocol.
Time Frame: up 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Split Dose R-CHOP
Number analyzed (Participants) | 26
proportion of participants | 0.346

5. Secondary Outcome: Summary of Treatment Emergent Serious Adverse Events by Grade and Organ System
Description: The incidence of serious adverse events will be reported for all subjects who received at least one dose of the study treatment.
Time Frame: up 6 months
Measure: Count of Units; unit: serious adverse events
Units Other Than Participants: serious adverse events
Groups:
- Grade 2: Moderate symptoms
- Grade 3: Severe symptoms
- Grade 4: Life-threatening symptoms
- Grade 5: Fatal
Arm/Group | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 26 | 26 | 26 | 26
Number analyzed (serious adverse events) | 2 | 30 | 7 | 3
serious adverse events
  Blood and lymphatic system disorders | 0 | 2 | 1 | 0
  Cardiac system disorders | 0 | 1 | 3 | 0
  Gastrointestinal disorders | 0 | 3 | 1 | 0
  General disorders and administration site conditions | 0 | 5 | 0 | 1
  Hepatobiliary disorders | 1 | 1 | 0 | 0
  Infections and infestations | 0 | 8 | 1 | 2
  Injury, poisoning and procedural complications | 0 | 3 | 0 | 0
  Metabolism and nutrition disorders | 1 | 1 | 1 | 0
  Nervous system disorders | 0 | 2 | 0 | 0
  Renal and urinary disorders | 0 | 1 | 0 | 0
  Skin and subcutaneous tissue disorders | 0 | 2 | 0 | 0
  Vascular disorders | 0 | 1 | 0 | 0

6. Secondary Outcome: Cancer-Specific Geriatric Assessment
Description: Cancer-specific geriatric assessment prior to, during, and after completion of chemotherapy treatments to evaluate for changes in physical function, mental health, cognition, and other relevant geriatric specific outcomes. The geriatric assessment measures will be summarized descriptively at each measurement time-point using appropriate descriptive statistics such as frequencies and percentages with standard errors for categorical variables, mean with standard error or median with quartiles for continuous variables.
Time Frame: up to 2 years 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Data collected up to approximately 6 months
Description: All-cause mortality is reported for all participants enrolled (N=27).
  Per protocol section 7.4.4: The incidence of serious adverse events will be reported for all subjects who received at least one dose of the study treatment (N=26).
  Per protocol section 8.3: Adverse events will be recorded from the beginning of informed consent until 2 weeks after completion of the last cycle of chemotherapy (N=27).
Arm/Group | Split Dose R-CHOP
All-Cause Mortality (participants affected / at risk) | 7/27
Serious Adverse Events (participants affected / at risk) | 9/26
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Split Dose R-CHOP (N=26)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorder, unknown (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fluid Volume Overload (General disorders) | 2 (4) — General disorders and administration site conditions
Cholecystitis (Hepatobiliary disorders) | 2 (2)
COVID-19 (Infections and infestations) | 3 (4)
Lung infection (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
LE blisters (Skin and subcutaneous tissue disorders) | 1 (2)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Split Dose R-CHOP (N=27)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (8)
Alanine aminotransferase increased (Investigations) | 6 (13)
Alkaline phosphatase increased (Investigations) | 10 (28)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 19 (66)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (General disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 9 (16)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood bicarbonate decreased (Investigations) | 3 (4)
Blood bilirubin increased (Investigations) | 5 (6)
Blood lactate dehydrogenase increased (Investigations) | 11 (25)
Blurred vision (Eye disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (4)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (2)
Chills (General disorders) | 4 (8)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (5)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Creatinine increased (Investigations) | 6 (16)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Delirium (Psychiatric disorders) | 2 (3)
Dental caries (Gastrointestinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (12)
Dizziness (Nervous system disorders) | 10 (17)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Edema limbs (General disorders) | 14 (25)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2)
Esophageal perforation (Gastrointestinal disorders) | 1 (1)
Keratitis sicca (Eye disorders) | 1 (1)
Pseudophakia (Eye disorders) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Eye pain (Eye disorders) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 6 (10)
Fatigue (General disorders) | 15 (29)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Fecal incontinence (Gastrointestinal disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Sore on lip (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 1 (1)
R sided maxillary pressure (Gastrointestinal disorders) | 1 (1)
Numbness of left foot and hand (General disorders) | 1 (1)
Stiffness in legs (in AM) (General disorders) | 1 (1)
Fluid Volume Overload (General disorders) | 2 (3)
Swollen Thumb (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (7)
GGT increased (Investigations) | 2 (2)
Glaucoma (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (13)
Heart failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (5)
Elevated LFTs (Hepatobiliary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot flashes (Vascular disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (13)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 10 (37)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (39)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (35)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 11 (31)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (15)
Hyponatremia (Metabolism and nutrition disorders) | 9 (28)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (18)
Hypotension (Vascular disorders) | 6 (11)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (8)
COVID-19 (Infections and infestations) | 4 (7)
Mild cold (Infections and infestations) | 1 (1)
Bacteruria (E. Coli) (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (3)
Small cut on leg (Injury, poisoning and procedural complications) | 1 (1)
Head pain (d/t syncope) (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 2 (3)
Deep tissue Injury (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
High chloride (Investigations) | 2 (4)
Low red count (Investigations) | 1 (3)
Low hematocrit (Investigations) | 1 (3)
Low monocytes (Investigations) | 1 (1)
Low creatinine (Investigations) | 1 (1)
Low uric acid (Investigations) | 1 (1)
Low MCH (Investigations) | 1 (1)
High RDW (Investigations) | 1 (1)
High neutrophils (Investigations) | 1 (2)
High monocytes (Investigations) | 1 (2)
Low globulin (Investigations) | 1 (1)
Low total protein (Investigations) | 2 (3)
High absolute immature granulocytes (Investigations) | 1 (1)
High myelocytes (Investigations) | 1 (1)
Low anion gap (Investigations) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Lethargy (Nervous system disorders) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Lung infection (Infections and infestations) | 4 (4)
Lymphocyte count decreased (Investigations) | 21 (103)
Malaise (General disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Multi-organ failure (General disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Bleeding Toe (Musculoskeletal and connective tissue disorders) | 1 (1)
stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocarditis (Cardiac disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Neutrophil count decreased (Investigations) | 12 (49)
Non-cardiac chest pain (General disorders) | 6 (6)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (10)
Paresthesia (Nervous system disorders) | 5 (10)
Paronychia (Infections and infestations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (16)
Phlebitis (Vascular disorders) | 2 (2)
Platelet count decreased (Investigations) | 14 (63)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (5)
Sinusitis (Infections and infestations) | 1 (1)
Scratched by dog (Skin and subcutaneous tissue disorders) | 1 (1)
Small flat blister-like spot on thigh (Skin and subcutaneous tissue disorders) | 1 (1)
wound buttocks & left foot (Skin and subcutaneous tissue disorders) | 1 (1)
bleeding wound on foot (Skin and subcutaneous tissue disorders) | 1 (1)
rash- macules, erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Broad actinic keratoses (Skin and subcutaneous tissue disorders) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Notalgia paresthetica (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
LE Blisters (Skin and subcutaneous tissue disorders) | 1 (3)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 3 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 6 (6)
Urinary incontinence (Renal and urinary disorders) | 6 (7)
Urinary retention (Renal and urinary disorders) | 3 (4)
Urinary tract infection (Infections and infestations) | 7 (9)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Vision decreased (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (16)
Vulval infection (Infections and infestations) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Weight gain (Investigations) | 2 (8)
Weight loss (Investigations) | 6 (14)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
White blood cell decreased (Investigations) | 14 (58)
Wound infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT03943901/Prot_SAP_000.pdf